CLINICAL TRIAL: NCT06844318
Title: Impact of Inflamatory Bowel Disease Activity on Frailty in Patients Over 60 Years
Brief Title: Impact of IBD Activity on Frailty in Patients Over 60 Years
Acronym: FRAGIL
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Other Study IDs: FRAGIL
Record Dates: First submitted 2025-02-03; First posted 2025-02-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: IBD
Keywords: eldearly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged ≥60 years with a diagnosis of IBD and clinical and/or biological disease activity: Patients aged ≥60 years with a diagnosis of inflamatory bowel disease (IBD) and clinical and/or biological disease activity

SUMMARY:
The goal of this observational, multicenter, descriptive, prospective, and longitudinal study is to evaluate the impact of IBD activity on frailty in a prospective and longitudinal cohort of patients with IBD, and also to assess the impact of frailty on the risk of hospitalization and mortality in patients with IBD aged ≥60 years.

The main questions it aims to answer are:

1. Can frailty and consequently the risk of complications (adverse events, hospitalization, and mortality) be reversed through proactive treatment in frail patients with active inflammatory bowel disease?
2. Which frailty index is the most effective for predicting the risk of complications in patients with active inflammatory bowel disease? At inclusion, clinical frailty indices will be calculated. Additionally, clinical variables related to IBD and comorbidities will be recorded. During follow ups visits frailty, comorbidities, IBD activity, changes in medical treatment for IBD, adverse effects, hospitalizations, and mortality will be reassessed.

DETAILED DESCRIPTION:
All consecutive patients meeting the selection criteria in the participating centres will be invited to participate.

-At inclusion, 4 clinical frailty indices (CFS-Clinical Frailty Scale, FRAGIL-VIG, Fried, VES-13) will be calculated. In addition, clinical variables on IBD (diagnosis, phenotype, extraintestinal manifestations, perianal disease, time of evolution of the disease, active treatments at the time of inclusion, treatment initiated, diagnostic tests available at the time of inclusion) and comorbidities (allowing calculation of the Charlson and Cumulative Illness Rating Scale for Geriatriscs [CIRS-G] indices) will be recorded.

Follow-up: a total of 3 follow-up visits will be conducted (at 3, 6 and 12 months) where frailty, comorbidities, IBD activity, changes in IBD medical treatment, adverse effects, hospitalisations and mortality will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥60 years with IBD (Crohn's disease or ulcerative colitis) diagnosed according to ECCO criteria and under follow-up in the IBD units of participating centers.
* Initiation of medical treatment (oral mesalazine, topical or systemic corticosteroids, immunosuppressants, and/or biologics) due to clinical activity based on PRO2 scales (UC: PRO >4; CD: PRO2 >14) and/or biological activity (fecal calprotectin ≥500 mg/kg, C-reactive protein ≥10 mg/L).
* Signed informed consent for inclusion.

Exclusion Criteria:

* Lack or withdrawal of informed consent.
* Unclassified/indeterminate colitis.
* Change in medical treatment solely due to adverse events.
* Initiation of treatment only with salicylates and/or topical steroids for disease activity.
* Treatment intensification to manage disease activity.
* Patients with an ostomy.
* Comorbidities with a life expectancy of less than one year.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥60 years with a diagnosis of IBD and clinical and/or biological disease activity.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of inflamatory bowel disease (IBD) activity on frailty in a prospective and longitudinal cohort of patients with IBD. | 12 months
  The evaluation of the impact of IBD activity will be measured by Patient Reported outcomes 2 (PRO-2).
  IBD clinical activity measured by PRO-2 for Crohn's disease (CD) is composed by:
  CD-PRO2: number of liquid daily stools and abdominal pain (0=none; 1=low; 2= moderate; 3= severe).
  IBD clinical activity measured by PRO-2 for ulcerative colitis (UC) is composed of 2 parts:
  UC-PRO2: stool number respect basal (0 =normal, same as usual; 1 = 1-2 stools more than the usual; 2 = 3-4 stools more than the usual; 3 = 5 or more stools more than the usual) and rectal bleeding (0 = none; 1 = visible blood in fences at least in half of them; 2 = visible blood in fences > half of them or mores; 3 = only blood).
  Clinic-biological activity: PRO2>4 in UC; PRO2>14 in CD
To assess the impact of frailty on the risk of hospitalization and mortality in patients with IBD aged ≥60 years. | 12 months
  The assessment of the impact of frailty will be measured by Fried Index. Fried Index is composed by a sum up of 5 parts, that follows:
  Unintended weight loss (score 0-1), Self-reported fatigue (score 0-1), Creep speed (score 0-1), Low physical activity (score 0-1), Weakness (score 0-1),
  The result of the total score is: Frail 3-5 points, pre- frail 1-2 points, "fit" 0 points.

CONTACTS AND LOCATIONS:
Overall Officials: Margalida Calafat, MD, PhD, Principal Investigator — Spanish Working Group on Crohn's disease and ulcerative colitis (GETECCU)
Locations (33):
- Spain (33):
  - Hospital Universitario Araba, Vitoria-Gasteiz, Alava
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Althaia Manresa, Manresa, Barcelona
  - Hospital del Mataró, Mataró, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Viladecans, Viladecans, Barcelona
  - Hospital Sierrallana de Torrelavega, Torrelavega, Cantabria
  - Hospital de Toledo, Toledo, Castille-La Mancha
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital de Henares, San Sebastián de los Reyes, Madrid
  - Hospital San Agustín de Avilés, Avilés, Principality of Asturias
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Astúrias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Dr Balmis, Alicante, Valencia
  - Hospital Denia, Denia, Valencia
  - Hospital Royo Villanova, San Gregorio, Zaragoza
  - Complejo Asistencial de Ávila, Ávila
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitari Dr Josep Trueta, Girona
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Ntra. Sra. de Candelaria, Santa Cruz de Tenerife
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario de la Fe, Valencia
  - Hospital Lozano Blesa, Zaragoza